CLINICAL TRIAL: NCT02822053
Title: Effectivity and Safety of Ultrasound-guided Percutaneously Laser Ablation for Refractory Neoplasms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-002
Record Dates: First submitted 2016-06-20; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Refractory Neoplasms
Keywords: Ultrasonography-guided Laser Ablation
MeSH Terms: conditions — Neoplasms

ARMS (1):
- US-guided laser ablation for refractory neoplasms (Experimental): The investigators used percutaneously US-guided laser ablation for patients with small hepatocellular carcinoma (single or multiple nodules of less than 3 cm in diameter), Child-Pugh A/B, PLT ≥ 50*10E9/L and PT ≤ 20s. Then the investigators estimated the safety and efficacy of this treatment through follow-up of US/CEUS/CT/MRI and the tumor markers every three months.
  Interventions: Procedure: US-guided laser ablation for refractory neoplasms

INTERVENTIONS:
Procedure: US-guided laser ablation for refractory neoplasms

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ultrasonography (US) -guided laser ablation liver, kidney, pancreas, lung and retroperitoneal tumors, the investigators used preoperative and postoperative US/CEUS/CT/MRI to assess lesions, and laboratory tests including the tumor markers to evaluate the general condition of patients. Intraoperative US/CEUS/CT would be applied to monitor ablation lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with small hepatocellular carcinoma (single or multiple nodules of less than 3 cm in diameter),
* Patients with Child-Pugh A/B,
* Patients with PLT ≥ 50*10E9/L and PT ≤ 20s.

Exclusion Criteria:

* Patients with blood coagulation dysfunction, ChildPugh ≥3, severe cardiopulmonary disease, intolerant anesthesia and upper gastrointestinal bleeding in shock.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
100 patients of refractory neoplasms with image-guided laser ablation-related effectivity as assessed by MRI | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Francica G, Petrolati A, Di Stasio E, Pacella S, Stasi R, Pacella CM. Influence of ablative margin on local tumor progression and survival in patients with HCC </=4 cm after laser ablation. Acta Radiol. 2012 May 1;53(4):394-400. doi: 10.1258/ar.2012.110471. Epub 2012 Mar 5. PMID 22393158
- [Result] Wu X, Zhou P, Ma S, Tian S, Deng J, Zhao Y. [Ultrasound-guided laser thermal ablation for treatment of small liver cancer at high-risk sites]. Nan Fang Yi Ke Da Xue Xue Bao. 2016 Jan;36(1):120-5. Chinese. PMID 26806751
- [Result] Di Costanzo GG, D'Adamo G, Tortora R, Zanfardino F, Mattera S, Francica G, Pacella CM. A novel needle guide system to perform percutaneous laser ablation of liver tumors using the multifiber technique. Acta Radiol. 2013 Oct;54(8):876-81. doi: 10.1177/0284185113489825. Epub 2013 May 23. PMID 23761559
- [Result] Zou X, Liu Q, Zhou X, He G, Yu M, Han Z, Meng X, Su H. Ultrasound-guided percutaneous laser and ethanol ablation of rabbit VX2 liver tumors. Acta Radiol. 2013 Mar 1;54(2):181-7. doi: 10.1258/ar.2012.110723. PMID 23482351
- [Result] Clements LW, Collins JA, Weis JA, Simpson AL, Adams LB, Jarnagin WR, Miga MI. Evaluation of model-based deformation correction in image-guided liver surgery via tracked intraoperative ultrasound. J Med Imaging (Bellingham). 2016 Jan;3(1):015003. doi: 10.1117/1.JMI.3.1.015003. Epub 2016 Mar 23. PMID 27081664
- [Derived] Jiang T, Deng Z, Tian G, Chen F, Bao H, Li J, Wang W. Percutaneous laser ablation: a new contribution to unresectable high-risk metastatic retroperitoneal lesions? Oncotarget. 2017 Jan 10;8(2):2413-2422. doi: 10.18632/oncotarget.13897. PMID 27974691